CLINICAL TRIAL: NCT00853710
Title: Validation of a Semiquantitative Screening Assay for PSA
Brief Title: Test Semiquantitative Prostate Specific Antigen (PSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-A01497-48; CRH 08/459/MN
Record Dates: First submitted 2009-02-24; First posted 2009-03-02 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Prostatic Diseases
Keywords: Prostate-Specific Antigen; Prostate Cancer; Cancer; Assay
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases; Neoplasms | interventions — Prostate-Specific Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rapid PSA assay on whole blood (Experimental)
  Interventions: Other: PSA assay

INTERVENTIONS:
Other: PSA assay — rapid prostate specific antigen assay.

SUMMARY:
The aim of the study is to compare the diagnostic performances of a simple and rapid PSA assay on whole blood to the standard plasma PSA assay.

DETAILED DESCRIPTION:
Screening and surveillance of prostate cancer typically involves sensitive laboratory techniques for the quantification of plasma prostate specific antigen (PSA). In this study, we determine the sensitivity and specificity of a simple test strip based PSA assay using only a few drops of whole blood as compared to a standard plasma PSA assay. Blood samples will be taken from hundred patients who are followed for a prostatic disease needing PSA surveillance. Before decantation of the samples, a few drops of blood will serve for the rapid test on strips. Plasma PSA levels will be determined with the TRACE ("Time Resolved Amplified Cryptate Emission") technology in homogeneous liquid phase. The results from the rapid test can then be compared to the plasma levels obtained by TRACE.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for prostate cancer or symptomatic benign prostatic disease, and for who a PSA assay is indicated.
* Patients must have given informed consent.

Exclusion Criteria:

* Patients followed for a disease other than prostatic.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Determination of the sensitivity and specificity of the rapid PSA assay by comparing the results obtained from the test strip reading by three independent blinded observers with those from standard plasma PSA assay. | day of test

SECONDARY OUTCOMES:
Determination of the threshold which maximizes the performance of the semiquantitative test. Determination of interobserver agreement. | at the last inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Dominique BELLET, Pr, Principal Investigator — Institut Curie
Locations (1):
- Centre Rene Huguenin, Saint-Cloud, France